CLINICAL TRIAL: NCT06870058
Title: A Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose of Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of NH280105 in Healthy Adult Participants
Brief Title: A Study of NH280105 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Nhwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NH280105-101
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NH280105-SAD (Experimental): SAD: Participants will either receive NH280105 or placebo across 4 cohorts
  * Cohorts 1, 2 and 4: Single dose on Day 1.
  * Cohort 3: Single dose on Days 1 and 15.
  Interventions: Drug: NH280105- SAD; Drug: Placebo
- NH280105- MAD (Experimental): MAD: Participants will receive either NH280105 or placebo, once daily for 14 days across 2-3 cohorts.
  Interventions: Drug: NH280105- MAD; Drug: Placebo

INTERVENTIONS:
Drug: NH280105- SAD — Dose formulation: Capsule Route of administration: oral
  Arms: NH280105-SAD
Drug: NH280105- MAD — Dose formulation: Capsule Route of administration: oral
  Arms: NH280105- MAD
Drug: Placebo — Matching placebo comparator

SUMMARY:
This is a Phase 1, randomized, double-blinded, placebo-controlled, single ascending dose (SAD) and multiple ascending dose (MAD) study to assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of NH280105 in healthy volunteers. In addition, this study will evaluate the effects of food on NH280105 under a two-period study setting.

DETAILED DESCRIPTION:
This study will be conducted in 2 parts: Part 1 (SAD) and Part 2 (MAD). Approximately 48 participants will be enrolled.

* Part 1 (Cohorts 1, 2, and 4): The study design includes a double-blind, placebo-controlled setting for SAD cohorts.
* Part 1 (Cohort 3): This cohort will be a double-blind, placebo-controlled, two-conditions (ie, fed vs. fasted), two-period, crossover setting for the Food-effect Cohort.
* Part 2: The study design includes a double-blind, placebo-controlled setting for MAD cohorts.

Oversight will be provided by a Safety Review Committee (SRC). Safety, tolerability, and PK/PD data (if available) of the preceding dose levels in both Part 1 (SAD) and Part 2 (MAD) will be reviewed by the SRC for dose escalation and the actual doses to be administered may be adjusted accordingly.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years at the time of informed consent.
2. At the discretion of the PI or designee, in good general health, with no significant medical history, and have no clinically significant abnormalities on physical examination at Screening and/or before the first administration of IP.
3. Body mass index (BMI) between ≥ 18.0 and ≤ 32.0 kg/m2 and weight ≥ 50 kg.
4. Clinical laboratory values within normal range as specified by the testing laboratory, unless deemed not clinically significant by the PI or designee.
5. Not pregnant or breastfeeding, or willing to cease breastfeeding.
6. Woman of childbearing potential or fertile man agrees to use an acceptable method of contraception from the start of Screening until 90 days after the last dose of IP. Acceptable methods of contraception are defined in protocol.

   Notes:
   1. Males must be surgically sterile (> 30 days since vasectomy with no viable sperm) or, if engaged in sexual relations with a WOCBP, must agree to use an acceptable contraceptive method.
   2. Females or males with same-sex partners (abstinence from penile-vaginal intercourse) or who are abstinent from heterosexual intercourse are not required to use contraception when this is their preferred and usual lifestyle.
   3. Males must not donate sperm from the first dose of IP until at least 90 days after the last dose of IP.
7. Able and willing to attend the necessary visits to the study site.
8. Able and willing to provide written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures.

Exclusion Criteria:

1. Use of tobacco or nicotine products exceeding 5 cigarettes (or equivalent) per week in any form within 30 days prior to IP administration on Day 1, or unwillingness to refrain from smoking, vaping, or using any nicotine products for at least 96 hours before the first IP administration, the onfinement period, and any Follow-up Visits.
2. Underlying physical or psychological medical condition that, in the opinion of the PI or designee, would make the participant unlikely to comply with the protocol or complete the study per protocol.
3. Blood or plasma donation or had significant blood loss (400 mL) within 30 days prior to the first administration of IP.
4. Fever (body temperature > 37.5°C) or symptomatic viral or bacterial infection within 2 weeks prior to Screening.
5. Infections requiring parenteral antibiotics within 6 months prior to Screening.
6. Positive test for hepatitis C antibody (HCV), hepatitis B surface antigen (HBsAg), human immunodeficiency virus (HIV) antibody.
7. Positive pregnancy test at Screening and/or on Day -1.
8. History of life-threatening infection (eg, meningitis).
9. Receiving live vaccine within 30 days prior to IP administration on Day 1 or require receiving live vaccination during the study or within 30 days end of the study.
10. Poor pill swallowing ability / poor venous access.
11. History of severe allergic or anaphylactic reactions, or sensitivity to the IP or its constituents; exceptions might be granted on a case-by-case basis upon agreement of the PI and the Sponsor.
12. History of malignancy, except for non-melanoma skin cancer, excised more than 2 years ago and cervical intraepithelial neoplasia that has been successfully cured more than 5 years prior to Screening.
13. Abnormal cardiac conditions and/or ECG findings at Screening

    * The Fridericia algorithm corrected QT interval (QTcF) of ECG during Screening Period is > 450 msec for males and > 470 msec for females or is considered abnormal with clinical significance as determined by the PI or designee.
    * Sustained (ie, 3 independent measurements within 30 minutes) heart rate (HR) > 100 or < 45 bpm.
    * Personal and/or family history of congenital long QT syndrome or sudden cardiac death.
14. BP is greater than 140/90 mmHg or below 90/40 mmHg and are considered by the PI/designee to be clinically significant.
15. History immunological disorders, auto-immune disorders, acquired or congenital immune deficiency, including autoimmune rheumatic disease.

    Note: participants with mild asthma controlled with occasional rescue inhaler only (no chronic therapy; no inhaled corticosteroids), and mild atopic dermatitis controlled with topic emollients only (no topical corticosteroids) are not excluded.
16. Exposure to any drugs that cause significant immunosuppression (including experimental therapies as part of a clinical study) within 4 months or 5 elimination half-lives (whichever is longer), prior to Screening.
17. Clinically significant abnormalities in laboratory test, including, including alkaline phosphatase (ALP), aspartate aminotransferase (AST), and alanine aminotransferase (ALT) > 1.5 × upper limit of normal (ULN) at Screening. Repeat testing at Screening is acceptable for out-of-range values following approval by the PI/designee.
18. Positive toxicology screening panel (urine test including qualitative identification of methamphetamine, opiates, cocaine, tetrahydrocannabinol (THC), pphencyclidine, benzodiazepines, barbiturates, methadone, tricyclic antidepressants (TCAs), amphetamine), nicotine (NB: positive nicotine is only exclusionary on Day -1, not during the screening period leading up to Day -1), and/or alcohol breath test at Screening or Day -1.
19. History of substance abuse or dependency or history of recreational IV drug use over the last 12 months (by self-declaration).
20. Regular alcohol consumption defined as > 10 standard drinks per week (where 1 standard drink = 360 mL of beer, 45 mL of 40% spirit or a 150 mL glass of wine) or > 4 standard drinks on any single day.
21. Unwilling to refrain from alcohol, methylxanthines, poppy seeds, and caffeine and caffeine consumption starting 48 hours before admission to the study site, throughout the confinement period, and for 48 hours prior to sequential dosing and any Follow-up Visits.
22. Use of any investigational medical device or investigational drug within 30 days or 5 half-lives of the investigational drug (whichever is longer) prior to the first administration of the IP.
23. Use of (or anticipated use of) any prescription drugs (other than hormonal contraception; oral contraceptive pills, long-acting implantable hormones, injectable hormones, a vaginal ring, or an intrauterine device [IUD]) within 30 days, OTC medication, nonsteroidal anti-inflammatory drug (NSAID), herbal remedies, supplements or vitamins within 14 days or 5 elimination half-lives (whichever is longer) prior to the first administration of IP and during the course of the study without prior approval of the PI and Sponsor MM. Simple analgesia (paracetamol) or other agents may be permitted at the discretion of the PI. Exception: Women of childbearing potential (WOCBP) are permitted to use hormonal contraception.
24. Unwilling to refrain from strenuous exercise (including weightlifting) from 48 hours prior to admission to the study site and from 48 hours prior to any Follow-up Visits.
25. Is or has an immediate family member (eg, spouse, parent/legal guardian, sibling, or child) who is investigational site or Sponsor staff directly involved with this study.
26. Anything that the PI considers would jeopardize the safety of the participant, prevent complete participation in the study, or compromise interpretation of study data.
27. Consumption of any known liver enzyme inducers or inhibitors, including foods or beverages such as citrus fruits (eg, tangerines, grapefruits, sweet oranges, limes, kumquats, citrons, oranges, lemons, etc.) and their juices, is prohibited within 7 days prior to the first administration of the IP.
28. Any major surgery within 6 months before Screening, or plan to have a surgery during the study. Participants meeting the following criterion are excluded from Part 1 - Cohort 3 (Food-effect Cohort).
29. Inability or unwillingness to consume a standard high-fat meal, as described in FDA Guidance for fed vs. fasted PK studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events following single and multiple adminstration of NH280105 | SAD- Up to Day 8; SAD FE- Up to Day 22; MAD- Up to Day 21 post first dose administration
Number of participants with change in laboratory parameters following treatment administration. | SAD- Up to Day 8; SAD FE- Up to Day 22; MAD- Up to Day 21 post first dose administration
  Hematology, clinical chemistry, coagulation and urinalysis will be assessed.
Number of participants with change in vital sign measurements following treatment adminstration | SAD- Up to Day 8; SAD FE- Up to Day 22; MAD- Up to Day 21 post first dose administration
  Blood pressure, heart rate, body temperature and respiratory rate will be assessed
Number of participants with change in physical examination following treatment administration | SAD- Up to Day 8; SAD FE- Up to Day 22; MAD- Up to Day 21 post first dose administration

SECONDARY OUTCOMES:
Plasma PK Parameters- Maximum plasma concentration (Cmax) for SAD and MAD cohorts | SAD- From Day 1 to Day 5; SAD FE- Day 1 to Day 5 and Day 15 to day 19; MAD- Day 1, Day2, Day3, Day 5, day 8, day 12, day 14, day 15, day 16, day 17and Day 18 post dose adminstration
Plasma PK Parameters-Time for maximum plasma concentration (Tmax) for SAD and MAD cohorts | SAD- From Day 1 to Day 5; SAD FE- Day 1 to Day 5 and Day 15 to day 19; MAD- Day 1, Day2, Day3, Day 5, day 8, day 12, day 14, day 15, day 16, day 17and Day 18 post dose adminstration
Plasma PK Parameters-Delay between the time of dosing and time of appearance of concentration (Tlag) for SAD and MAD cohorts | SAD- From Day 1 to Day 5; SAD FE- Day 1 to Day 5 and Day 15 to day 19; MAD- Day 1, Day2, Day3, Day 5, day 8, day 12, day 14, day 15, day 16, day 17and Day 18 post dose adminstration
Plasma PK Parameters-Area Under Curve for SAD and MAD cohorts | SAD- From Day 1 to Day 5; SAD FE- Day 1 to Day 5 and Day 15 to day 19; MAD- Day 1, Day2, Day3, Day 5, day 8, day 12, day 14, day 15, day 16, day 17and Day 18 post dose adminstration
Plasma PK Parameters-Elimination half-life (t1/2) for SAD and MAD cohorts | SAD- From Day 1 to Day 5; SAD FE- Day 1 to Day 5 and Day 15 to day 19; MAD- Day 1, Day2, Day3, Day 5, day 8, day 12, day 14, day 15, day 16, day 17and Day 18 post dose adminstration
Plasma PK Parameters- Elimination rate constant (Kel) for SAD and MAD cohorts | SAD- From Day 1 to Day 5; SAD FE- Day 1 to Day 5 and Day 15 to day 19; MAD- Day 1, Day2, Day3, Day 5, day 8, day 12, day 14, day 15, day 16, day 17and Day 18 post dose adminstration
Plasma PK Parameters-Volume of distribution (Vz/F) for SAD and MAD cohorts | SAD- From Day 1 to Day 5; SAD FE- Day 1 to Day 5 and Day 15 to day 19; MAD- Day 1, Day2, Day3, Day 5, day 8, day 12, day 14, day 15, day 16, day 17and Day 18 post dose adminstration
Plasma PK Parameters- Clearance per bioavailability (CL/F) for SAD and MAD cohorts | SAD- From Day 1 to Day 5; SAD FE- Day 1 to Day 5 and Day 15 to day 19; MAD- Day 1, Day2, Day3, Day 5, day 8, day 12, day 14, day 15, day 16, day 17and Day 18 post dose adminstration
Plasma PK Parameters- Mean Residence time (MRT) for SAD and MAD cohorts | SAD- From Day 1 to Day 5; SAD FE- Day 1 to Day 5 and Day 15 to day 19; MAD- Day 1, Day2, Day3, Day 5, day 8, day 12, day 14, day 15, day 16, day 17and Day 18 post dose adminstration
To evaluate the PD effect of repeated oral doses of NH280105 on the plasma Lp-PLA2 inhibition from baseline | SAD- From Day 1 to Day 5; SAD FE- Day 1 to Day 5 and Day 15 to day 19; MAD- Day 1, Day2, Day3, Day 5, day 8, day 12, day 14, day 15, day 16, day 17and Day 18 post dose adminstration
Plasma PK: The ratio of fed/fasted on Cmax- Maximum plasma concentration | Part 1 - Food effect Cohort (Cohort 3) From Day 1 to Day 19 except Day 14.
Plasma PK: The ratio of fed/fasted on AUC(0-t)- Area under curve from 0 to timepoint | Part 1 - Food effect Cohort (Cohort 3) From Day 1 to Day 19 except Day 14.
Plasma PK: The ratio of fed/fasted on AUC(0-inf)- Area under curve from 0 to infinity | Part 1 - Food effect Cohort (Cohort 3) From Day 1 to Day 19 except Day 14.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sun, Study Director — Head of Global BD
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No